CLINICAL TRIAL: NCT01101932
Title: A Phase 1, Placebo-Controlled, Multiple-Dose Escalation Trial Evaluating The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-04308515 (Part 1), And A Single Dose Pharmacokinetic Assessment Of A PF-04308515 Tablet Formulation (Part 2), In Healthy Volunteers
Brief Title: Multiple Dose Escalation Trial Of PF-04308515 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: B0861002
Record Dates: First submitted 2010-03-11; First posted 2010-04-12 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics/Pharmacodynamics; Rheumatoid Arthritis; healthy volunteers
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- (Part 1) PF-04308515 (Experimental)
  Interventions: Drug: PF-04308515
- (Part 1) Solution Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- (Part 2) PF-04308515 Tablet (Experimental)
  Interventions: Drug: PF-04308515 Tablet

INTERVENTIONS:
Drug: PF-04308515 — PF-04308515 will be provided as an oral solution administered at doses of 3, 10, 30 and 100 mg. If an optional cohort is needed the dose would not exceed the established toxicokinetic exposure limits. Solution will be administered orally once daily for 14 days.
  Arms: (Part 1) PF-04308515
Drug: Placebo — Placebo solution will be administered to those volunteers who are randomized to the placebo arm. Placebo solution will be administered orally once daily for 14 days.
  Arms: (Part 1) Solution Placebo
Drug: PF-04308515 Tablet — Tablet formulation to administer a 20 mg dose will be administered to volunteers in Part 2. The study medication will be administered orally once daily for 1 day.
  Arms: (Part 2) PF-04308515 Tablet

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics (how the drug effects certain target sites of activity in the body) of escalating doses of oral PF-04308515 in healthy volunteers for 14 days as well as one oral dose of a tablet formulation administered for 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 55 years, inclusive
* Healthy females between 18 and 44 years, inclusive
* Females are required to be surgically sterile

Exclusion Criteria:

* Evidence or history of clinically significant disease
* Post-menopausal women
* History of intolerance or significant adverse effects with glucocorticoid therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple doses of PF-04308515 as assessed by adverse event reporting, clinical laboratory results, vital signs, physical examinations and electrocardiograms (ECGs). | 14 days
Characterization of pharmacokinetic parameters of PF-04308515 after multiples doses which will include: Cmax, Tmax, AUC, CL/F, Vz/F, t1/2. Urinary excretion including AE% and CLr will be assessed at steady state. | 14 days
Change from baseline will be utilized to assess PF-04308515's pharmacodynamic effect on biochemical and metabolic biomarkers after 14 days of dosing. | 14 days
For the tablet pharmacokinetics:Cmax, Tmax, AUClast, AUCinf, CL/F, Vz/F, t1/2 will be calculated from the PF-04308515 plasma concentration versus time data. | 1 day
Safety and tolerability of 1 oral dose of a tablet formulation of PF-04308515 as assessed by adverse event reporting, clinical laboratory results, vital signs, physical examinations and electrocardiograms (ECGs). | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0861002&StudyName=Multiple%20Dose%20Escalation%20Trial%20Of%20PF-04308515%20In%20Healthy%20Volunteers